CLINICAL TRIAL: NCT00005658
Title: Childhood Onset Psychotic Disorders: An Open Trial With the Amino Acid Glycine
Brief Title: Glycine to Treat Psychotic Disorders in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000122; 00-M-0122
Record Dates: First submitted 2000-05-09; First posted 2000-05-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Psychotic Disorder; Schizoaffecitve Disorder; Schizophrenia
Keywords: Biochemical; Schizophrenia; NMDA; Adolescence; Psychosis; Child Psychosis; Biochemical Correlates; Brain Imaging; Glycine; Adjunctive Glycine Therapy
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Glycine

INTERVENTIONS:
Drug: Glycine

SUMMARY:
This study will test the safety and effectiveness of the amino acid glycine in treating psychotic disorders in children. The drug will be given as an adjunct (in addition) to the patient's current antipsychotic medication.

Children age nine to 18 with schizophrenia or schizoaffective disorder whose symptoms began before age 13 may be eligible for this 10-week study. Patients will be hospitalized during the course of the trial. Weekend visits home may be permitted.

Children enrolled in the study will be evaluated during a two-week pre-treatment period with written tests for IQ and academic functioning and with a magnetic resonance imaging (MRI) scan of the brain. For the MRI, the child lies on a table that slides into a large donut-shaped machine with a strong magnetic field. This procedure produces images of the brain that may help identify brain abnormalities in schizophrenia that develop in childhood.

During the eight-week treatment phase, patients will receive glycine powder dissolved in water once a day, in addition to their other antipsychotic medications. They will undergo the following additional procedures during the course of treatment:

1. Comprehensive psychiatric examination
2. Blood pressure and pulse monitoring once a week
3. Blood tests every other week - About one ounce of blood is drawn per week to measure glycine levels
4. Eye movement study at week eight - Using a technique called infrared oculography, special detectors measure infrared light reflected off the child's eyes while he or she watches a moving square on a video monitor.
5. Lumbar puncture (spinal tap) once during the study - About one-half ounce of cerebrospinal fluid (the fluid surrounding the brain and spinal cord) is withdrawn through a needle placed in the lower part of the spine for analysis of brain chemicals.

Patients who respond well may continue to receive glycine treatment through their referring physician after the study is completed.

NIMH will follow patients by phone every six months and with visits at two-year intervals.

DETAILED DESCRIPTION:
The ability of glycine to potentiate the NMDA receptor-complex, along with the fact that it is well tolerated in short-and long-term administration, has raised the possibility that it may provide an effective treatment of augmentation for neuroleptic-resistant negative symptoms of schizophrenia. Up to ten children and adolescents, ages 9-18, meeting DSM-IV criteria for schizophrenia, schizoaffective disorder and psychotic disorder not otherwise specified with onset of psychosis by age 12 who have failed at least two prior antipsychotics entering this protocol on their current antipsychotic medication(s) will participate in an open 8-week trial of adjunctive glycine therapy. In addition to the potential benefits, if glycine therapy ameliorates enduring negative symptoms of schizophrenia, we anticipate that recruiting these rare patients will be facilitated by the availability of this new treatment.

This study will provide pilot data regarding the beneficial effects and safety of adjunctive glycine therapy for children and adolescents with treatment refractory psychotic disorders. The availability of newer alternate treatments is also important for recruitment of patients in the broader study of the neurobiology and genetics of very early onset schizophrenia.

Children and adolescents ages nine to eighteen will be allowed into the study. Subjects entering the protocol as new patients will be characterized by clinical phenomenology, eye tracking, MRI brain imaging, cerebrospinal fluid, plasma and urinary biochemistry, and chromosomal analysis. Patients with prominent mood symptoms who have required the addition of mood stabilizing agents such as lithium or valproic acid will be allowed to remain on these medications for the duration of the treatment trial, if clinically indicated. Liver chemistries will be checked at baseline and at the end of the study.

All first-degree relatives are interviewed in person and undergo eye tracking measurement and contribute blood cell lines as part of a genetic study of the cohort (84-M-0050).

ELIGIBILITY:
Patients with their psychosis in a moderate to severe range defined as a SANS score of 5 or above, a SAPS score of 5 or above and/or a BPRS score of 30 or above.

Males and females, age 9-18 meeting DSM-IV criteria for schizophrenia, schizoaffective disorder or psychotic disorder not otherwise specified with onset of psychosis before their 13th birthday.

Patients must have had their 9th birthday by the end of drug washout.

Patients with failure of two prior antipsychotic treatments, or discontinuation of effective clozapine or olanzapine treatment due to intolerable side effects.

Patients with a premorbid IQ test less than 70.

No patients with any significant neurological/medical disorder; and/or active alcohol or drug abuse.

No patients judged to be at serious suicidal risk.

Females who are physically capable of pregnancy must agree to avoid pregnancy throughout the study. Should pregnancy occur during the study, the patient will be unable to continue.

MRI exam will not be given to patients with any metal prostheses, surgical clips, or other metal implants, or cannot tolerate the procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10
Dates: Start 2000-05; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ambrosini PJ, Metz C, Prabucki K, Lee JC. Videotape reliability of the third revised edition of the K-SADS. J Am Acad Child Adolesc Psychiatry. 1989 Sep;28(5):723-8. doi: 10.1097/00004583-198909000-00013. PMID 2793800
- [Background] Alaghband-Rad J, McKenna K, Gordon CT, Albus KE, Hamburger SD, Rumsey JM, Frazier JA, Lenane MC, Rapoport JL. Childhood-onset schizophrenia: the severity of premorbid course. J Am Acad Child Adolesc Psychiatry. 1995 Oct;34(10):1273-83. doi: 10.1097/00004583-199510000-00012. PMID 7592264
- [Background] Frazier JA, Giedd JN, Kaysen D, Albus K, Hamburger S, Alaghband-Rad J, Lenane MC, McKenna K, Breier A, Rapoport JL. Childhood-onset schizophrenia: brain MRI rescan after 2 years of clozapine maintenance treatment. Am J Psychiatry. 1996 Apr;153(4):564-6. doi: 10.1176/ajp.153.4.564. PMID 8599409